CLINICAL TRIAL: NCT02730832
Title: Validation of Scale to Evaluate the Perception of Oral Health in Patients With Schizophrenia
Brief Title: Validation of a Scale to Evaluate the Perception of Oral Health in Patients With Schizophrenia
Acronym: QUALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: DENIS 2015
Record Dates: First submitted 2016-03-21; First posted 2016-04-07 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with schizophrenia (Experimental)
  Interventions: Other: Questionnaires completed at D0; Other: Questionnaires completed at D15 (test-retest for 30 patients)

INTERVENTIONS:
Other: Questionnaires completed at D0
Other: Questionnaires completed at D15 (test-retest for 30 patients)

SUMMARY:
Apart from objective criteria for the evaluation of oral health (CAO, CPI…), there are no scales to evaluate the oral health of patients with schizophrenia. The only scales that do exist are for the population at large, children or the elderly. Given the severely deteriorated oral health in these schizophrenic populations, it is important to have a tool to evaluate their perception of the quality of their oral health so as to better orientate prevention programmes.

The aim of this study is to validate a tool to measure the perception of oral health in patients with schizophrenia.

To do this, patients will be invited to complete a series of self-questionnaires relative to the concept of oral health.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia according to DSM V
* Hospitalized patients or outpatients who have been taking an antipsychotic treatment for more than 2 years
* Patients older than 18 years
* Patients who have provided oral informed consent to take part in the study

Exclusion Criteria:

* Patients who are psychiatrically unstable or delusional
* Subjects on chemotherapy
* Adults under guardianship
* Patients without national health insurance cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Perception of oral health by OHIP-14 scales | At inclusion
Evaluation of quality of life by GOHAI scales | At inclusion
Mc Nair Memory Questionnaire | At inclusion
Evaluation of negative symptoms by scale | At inclusion
Beck Depression Scale | At inclusion
Evaluation of quality of life by S-Qol | At inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CH La Chartreuse, Dijon, France

REFERENCES:
- [Result] Siu-Paredes F, Rude N, Rat C, Reynaud M, Hamad M, Moussa-Badran S, Denis F. The Schizophrenia Coping Oral Health Profile. Development and Feasibility. Transl Neurosci. 2018 Jun 20;9:78-87. doi: 10.1515/tnsci-2018-0014. eCollection 2018. PMID 29967693
- [Derived] Frederic D, Corinne R, Matthieu R, Francesca SP, Stephanie TJ, Nathalie R. The Schizophrenia Oral Health Profile: Development and Feasibility. Transl Neurosci. 2018 Sep 22;9:123-131. doi: 10.1515/tnsci-2018-0019. eCollection 2018. PMID 30263228